CLINICAL TRIAL: NCT06032936
Title: An Open-label, Non-randomized, Multi-cohort, Multi-center Phase Ia/Ib Study Evaluating the Efficacy and Safety of BBP-398 in Combination With Osimertinib in Locally Advanced or Metastatic NSCLC Patients With EGFR Mutations
Brief Title: BBP-398 in Combination With Osimertinib in Locally Advanced or Metastatic NSCLC Patients With EGFR Mutations
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business reason
Sponsor: LianBio LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LB1002-102
Record Dates: First submitted 2023-07-31; First posted 2023-09-13 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: NSCLC
MeSH Terms: interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BBP-398 + Osimertinib (Experimental): Phase Ia (Dose Escalation):
  Dose level 1: (starting dose level) The one lower dose level than RP2D of BBP-398 monotherapy in Chinese patients (RP2D -1) with Osimertinib 80 mg Dose level 2: RP2D The same dose level to RP2D of BBP-398 monotherapy in Chinese patients with Osimertinib 80 mg Note: The dosing interval and regimen might be changed based on emerging data of Study NAV-1001, LB1002-101 and this study. The proposed new dosing regimen will be submitted in a memo to EC for approval before execution.
  Phase Ib (Efficacy Expansion):
  Osimertinib 80mg QD + BBP-398 RP2D QD
  Interventions: Drug: BBP-398; Drug: osimertinib

INTERVENTIONS:
Drug: BBP-398 — BBP-398 (formerly known as IACS-15509) is a potent, selective, orally active allosteric inhibitor of SHP2, a tyrosine phosphatase that plays a key role in the RTK -MAPK signal transduction pathway. Key components of the MAPK pathway include the small GTPase RAS, the serine/threonine-protein kinase RAF, mitogen-activated protein kinase (MEK) and ERK. In cells, SHP2 binds to phosphorylated tyrosine residues in the intracellular domain of RTKs such as the EGFR, leading to activation of the downstream MAPK signaling pathway.
  Other Names: IACS-15509
Drug: osimertinib — Osimertinib is a mutant-selective, third-generation EGFR inhibitor that targets both EGFR-activating mutations (e.g., exon 19 deletion and L858R) and EGFR-dependent on-target resistance mutation toward the 1st generation EGFR inhibitor (i.e., T790M). It is currently a first-line therapy for EGFR-mutant (EGFRmut) NSCLC, with average progression-free survival of approximately 19 months in previously untreated subjects.

SUMMARY:
This is an open-label, non-randomized, multi-cohort, multi-center Phase Ia/Ib study for BBP-398 in combination with Osimertinib to evaluate the safety, tolerability, pharmacokinetics, determine MTD and/or RP2D, and anti-cancer activity in locally advanced or metastatic NSCLC patients with EGFR mutations and with previously 3rd generation EGFR-TKIs treated or EGFR-TKI-naive.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have the ability to understand and the willingness to sign a written informed consent document.
* Patients must be willing and able to comply with the scheduled visits, treatment plan, laboratory tests and other specified study procedures.
* Age ≥18, male or female.
* Patients are not suitable for surgical resection and must have histologically or cytologically confirmed advanced or metastatic NSCLC with documented EGFR sensitivity mutation (at any time since the initial diagnosis of NSCLC) to confirm susceptibility to EGFR-TKI therapy.
* Patients must have measurable disease by RECIST v1.1.
* ECOG performance status ≤2.
* Patients must have a life expectancy of ≥12 weeks as estimated at the time of screening.
* Patients must have adequate organ function.

Exclusion Criteria:

* Patients with a known additional malignancy that is progressing or requires active treatment.
* Patients who have previously received a SHP-2 inhibitor.
* Patients who are hypersensitivity to BBP-398/ Osimertinib or active or inactive excipients.
* Treatment with any of the following anti-cancer therapies prior to the first dose within the stated timeframes.
* Pregnant or breastfeeding female patients.
* Patients with untreated symptomatic brain metastases and/or meningeal metastases.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-07-27 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (TEAEs) | From the first study administration to approximately 28 days after the last study administration
  Incidence and severity of treatment-emergent adverse events (TEAEs).
Serious adverse events (SAEs) | Administration to approximately 28 days after the last study administration
  Incidence and severity of Serious adverse events (SAEs)
Phase Ib: ORR assessed by the investigator according to RECIST v1.1 | Every 8 weeks from first dose administration to the date of progression determined by the investigator or death due to any cause, whichever came first, assessed approximately 48 months.
  ORR is defined as number of patients with confirmed responses of CR or PR, divided by the total number of treated patients with measurable disease at baseline assessed by the investigator.

SECONDARY OUTCOMES:
Phase Ia: QT Interval | Approximately 6 months
  Evaluated by comparing the changes using electrocardiogram in the post-dose to the pre-dose.
Maximum plasma concentration (Cmax) | Approximately 6 months
  To characterize the pharmacokinetic parameter Maximum plasma concentration (Cmax) of BBP-398 and/or Osimertinib and its metabolites
Area under the plasma concentration versus time curve (AUC) | Approximately 6 months
  To characterize the pharmacokinetic parameter Area under the plasma concentration versus time curve (AUC) of BBP-398 and/or Osimertinib and its metabolites
Time to Reach Maximum Plasma Concentration (Tmax) | Approximately 6 months
  To characterize the pharmacokinetic parameter time to reach maximum plasma concentration (Tmax) of BBP-398 and/or Osimertinib and its metabolites.
Apparent total plasma clearance (CL/F) | Approximately 6 months
  To characterize the pharmacokinetic parameter Apparent total plasma clearance (CL/F) of BBP-398 and/or Osimertinib and its metabolites.
Terminal elimination half-life (t1/2) | Approximately 6 months
  To characterize the pharmacokinetic parameter Terminal elimination half-life (t1/2) of BBP-398 and/or Osimertinib and its metabolites.
Accumulation ratio (Racc) | Approximately 6 months
  To characterize the pharmacokinetic parameter Accumulation ratio (Racc) of BBP-398 and/or Osimertinib and its metabolites.
Phase Ib: DOR | Every 8 weeks from first evaluation as CR or PR to the first evaluation as PD or death of any cause, whichever came first, assessed approximately 24 months.
  DOR assessed by the investigator according to RECIST v1.1. DoR is defined as time interval from the first evaluation as CR or PR to the first evaluation as PD or death of any cause assessed by the investigator (percent of patients with ≥6 months, ≥9 months, and ≥12 months DoR will be reported).
Phase Ib: PFS | Every 8 weeks from first evaluation as CR or PR to the first evaluation as PD or death of any cause, whichever came first, assessed approximately 24 months.
  PFS assessed by the investigator according to RECIST v1.1. PFS is defined from the first date of treatment to the date of progression determined by the investigator or death due to any cause (only for dose expansion).
Phase Ib: OS | From the first date of treatment until date of death, assessed approximately 48 months.
  including 1-year and 2-years survival rate. OS is defined from the first date of treatment until date of death (only for dose expansion).

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Master, Principal Investigator — Sun Yat-sen University
Locations (5):
- China (5):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guanzhou, Guangdong
  - Jilin Cancer Hospital, Changchun, Jilin
  - Shandong Cancer Hospital, Jinan, Shandong
  - West China Hospital Sichuan University, Chengdu, Sichuan